CLINICAL TRIAL: NCT06287450
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Respiratory Syncytial Virus IN006 Bivalent mRNA Vaccine (IN006) in Healthy Adult Participants
Brief Title: A Study to Describe the Safety and Immunogenicity of a Respiratory Syncytial Virus Vaccine IN006 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Shenxin Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN006001
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: mRNA Vaccine; IN006; Respiratory syncytial virus; Viral Diseases; Messenger RNA; Innorna; Shenxin; Vaccines; Respiratory tract infections; Safety; Reactogenicity; Immunogenicity; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Dose A in Younger Adults (Experimental): Single injection of Dose A of IN006 or matching-placebo on Day 0.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 2: Dose B in Younger Adults (Experimental): Single injection of Dose B of IN006 or matching-placebo on Day 0.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 3: Dose C in Younger Adults (Experimental): Single injection of Dose C of IN006 or matching-placebo on Day 0.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 4: Dose D in Younger Adults (Experimental): Single injection of Dose D of IN006 or matching-placebo on Day 0.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 5: Dose B in Older Adults (Experimental): One injection of either Dose B of IN006 or matching-placebo on Day 0. Participants who initially assigned to receive IN006 on Day 0 will be further randomized to receive a second injection of either IN006 or matching-placebo approximately 12 months later.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 6: Dose C in Older Adults (Experimental): One injection of either Dose C of IN006 or matching-placebo on Day 0. Participants who initially assigned to receive IN006 on Day 0 will be further randomized to receive a second injection of either IN006 or matching-placebo approximately 12 months later.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo
- Cohort 7: Dose D in Older Adults (Experimental): One injection of either Dose D of IN006 or matching-placebo on Day 0. Participants who initially assigned to receive IN006 on Day 0 will be further randomized to receive a second injection of either IN006 or matching-placebo approximately 12 months later.
  Interventions: Biological: Bivalent RSV Vaccine (IN006); Biological: Placebo

INTERVENTIONS:
Biological: Bivalent RSV Vaccine (IN006) — Formulation for injection
Biological: Placebo — 0.9% sodium chloride (normal saline) injection

SUMMARY:
The study will evaluate the safety, tolerability, and immunogenicity of a single injection of up to 4 dose levels of IN006 in younger adults and 3 dose levels of IN006 in older adults; of a revaccination of IN006 given approximately 12 months after the initial vaccination in older adults.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female participants aged ≥18 to 59 years of age (Part 1) or ≥ 60 to 79 years of age (Part 2).
2. Body weight ≥ 50 kg for males and ≥ 45 kg for females and body mass index (BMI) in the range of 18.5 to 35 kg/m^2.
3. For all women of childbearing potential (WOCBP) females must be non-pregnant and non-lactating and must use an appropriate contraceptive method from at least 30 days prior to study vaccination (an effective contraception) until at least 6 months after study vaccination. Women not of childbearing potential must be postmenopausal for ≥ 12 months.
4. Male participants who are non-sterilized and sexually active must be willing to use an acceptable, effective contraceptive method from at least 30 days prior to study vaccination until at least 6 months after study vaccination.
5. Able and willing to complete the study procedures during the entire study Follow-up period.
6. Can understand the study procedures, voluntarily sign the informed consent form after informed consent, and be able to comply with the requirements of the clinical study protocol.

Key Exclusion Criteria:

1. Pregnant or lactating at Screening or prior to vaccination or planning to become pregnant (self or partner) at any time during the study, including the specified Follow-up period.
2. Participants with a known (documented or self-reported) history of Guillain-Barré syndrome, encephalomyelitis, or transverse myelitis.
3. Participants with a known (documented or self-reported) history of heart disease (eg, heart failure, recent coronary artery disease, myocarditis, pericarditis, cardiomyopathy, or atrial fibrillation). Note: chronic stable coronary artery disease that is considered mild may be allowed at the discretion of the Investigator.
4. Participants with uncontrolled hypertension (supine systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg at Screening). Results at Screening may be confirmed by single repeat at the discretion of the Investigator.
5. Participants with a Screening 12-lead ECG following at least 5 minutes of supine rest demonstrating a Fridericia corrected QT (QTcF) interval > 450 msec (for males) or > 470 msec (for females) or a QRS interval ≥ 120 msec.
6. Participants with clinically significant abnormalities that indicate or meet the definition of a Grade 1 or greater abnormality for Part 1, or a Grade 2 or greater abnormality for Part 2 as delineated in the FDA guidance "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials".
7. Participants with acute medical or febrile illness (body temperature > 38.0°C or 100.4°F) within one day prior to vaccination.
8. History of severe hypersensitivity reactions, including anaphylaxis or other significant adverse reactions to any components of a mRNA vaccine or known components of IN006.
9. Received any live attenuated vaccines ≤ 28 days prior to vaccination or plans to receive any licensed vaccines within 28 days before the study vaccination, with the exception of licensed inactivated influenza vaccine or non-replicating influenza vaccine which may be given ≥ 14 days prior to the first study vaccination.
10. Received immunomodulatory, immunostimulatory, or immunosuppressant drugs including interferon and cytotoxic drugs within 90 days of Screening or planning to receive during the study.
11. Received a previous vaccination with any licensed or investigational RSV vaccine prior to enrollment or planned to receive at any time throughout the duration of the study.
12. Received immunoglobulin and/or any blood products within 120 days of vaccination.
13. Use of systemic corticosteroids exceeding the equivalent of 10 mg/day of prednisone for ≥ 10 days within 30 days of Screening or planning to receive during the study.
14. History of a known bleeding disorder that would, in the opinion of the Investigator, contraindicate intramuscular (IM) injection.
15. History of congenital or acquired immunodeficiency including HIV or immunosuppressive disorder, asplenia, or recurrent severe infections.
16. Known or suspected clinically significant or unstable significant hematologic (including clotting disorders), renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies and untreated seasonal allergies) that may interfere with the study evaluations or the participants ability to complete the study, in the opinion of the Investigator.
17. History of, or current positive results for, any of the following serological tests: HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCV Ab), or syphilis.
18. Recent history of major surgical procedures within 90 days of Screening.
19. Treatment with an investigational product within 30 days, or 5 half-lives (whichever is longer) preceding vaccination.
20. Blood donation of approximately 500 mL or more within 60 days prior to vaccination.
21. Any other reason to be excluded in the opinion of the Investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Solicited Local and Systemic Adverse Reactions Through 14 Days After Initial Vaccination | From initial vaccination up to14 days post initial vaccination
Percentage of Participants With Unsolicited Adverse Events (AEs) Through 28 Days After Initial Vaccination | From initial vaccination up to 28 days post initial vaccination
Percentage of Participants With Any Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), and AEs Leading to Study Discontinuation Through 12 Months After Initial Vaccination | From initial vaccination up to 12 months post initial vaccination
Percentage of Participants With Any Medically Attended AEs (MAAEs) Through 6 Months After Initial Vaccination | From initial vaccination up to 6 months post initial vaccination

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) for Neutralizing Antibodies Against RSV A and RSV B (Via Neutralization Assay) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
Geometric Mean Fold Rise (GMFR) for Neutralizing Antibodies Against RSV A and RSV B (Via Neutralization Assay) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
Vaccine Response Rate for Neutralizing Antibodies Against RSV A and RSV B (Via Neutralization Assay) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
GMC for Pre-F Specific Binding Antibodies Against RSV A and RSV B (Via Enzyme Immunoassay [EIA]) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
GMFR for Pre-F Specific Binding Antibodies Against RSV A and RSV B (Via Enzyme Immunoassay [EIA]) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
Vaccine Response Rate for Pre-F Specific Binding Antibodies Against RSV A and RSV B (Via Enzyme Immunoassay [EIA]) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
Frequency of Pre-F Specific IFN-γ/IL-4 Secreting T cells (Via Enzyme-Linked Immunospot [ELISpot] Assay) | Before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1, 3, 6 and 12 months post-initial vaccination (Part 2, participants aged 60 to 79 years)
Frequency of Pre-F Specific CD4 and CD8 T Cells Expressing Activation Markers (Via Intracellular Cytokine Staining [ICS] Assay) | Before vaccination, and 2 weeks and 1 month post-vaccination (Part 1, participants aged 18 to 59 years); before vaccination, and 2 weeks and 1 month post-initial vaccination (Part 2, participants aged 60 to 79 years)
Percentage of Participants (Part 2, Aged 60 to 79 Years) With Solicited Local and Systemic Adverse Reactions Through 14 Days After Revaccination | From second vaccination up to 14 days post revaccination
Percentage of Participants (Part 2, Aged 60 to 79 Years) With Unsolicited AEs Through 28 Days After Revaccination | From second vaccination up to 28 days post revaccination
Percentage of Participants (Part 2, Aged 60 to 79 Years) With Any MAAEs Through 6 Months After Revaccination | From second vaccination up to 6 months post revaccination
Percentage of Participants (Part 2, Aged 60 to 79 Years) With Any SAEs, AESIs, and AEs Leading to Study Discontinuation Through 6 Months After Revaccination | From second vaccination up to 6 months post-revaccination

IPD SHARING:
Plan to Share IPD: Undecided